CLINICAL TRIAL: NCT01070927
Title: An Exploratory Study on Anti-tumour Activity of Orally Administered RO4929097, a Gamma-secretase Inhibitor, as a Single Agent in Patients With Recurrent or Refractory Non-Small Cell Lung Cancer (NSCLC).
Brief Title: An Exploratory Study of RO4929097 in Patients With Recurrent or Refractory Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP22383; 2008-006384-37
Record Dates: First submitted 2010-02-16; First posted 2010-02-18 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Non-Squamous Non-Small Cell Lung Cancer
MeSH Terms: interventions — 2,2-dimethyl-N-(6-oxo-6,7-dihydro-5H-dibenzo(b,d)azepin-7-yl)-N'-(2,2,3,3,3-pentafluoropropyl)malonamide

ARMS (2):
- cohort 1 (Experimental)
  Interventions: Drug: RO4929097
- cohort 2 (Experimental)
  Interventions: Drug: RO4929097

INTERVENTIONS:
Drug: RO4929097 — 80mg po daily, 3 days on 4 days off schedule
  Arms: cohort 1
Drug: RO4929097 — recommended phaseII dose, orally once daily, 3 days on 4 days off schedule
  Arms: cohort 2

SUMMARY:
This study will evaluate the anti-tumour activity, safety and tolerability of RO4929097 as monotherapy in patients with recurrent or refractory non-small cell lung cancer. Patients will receive oral doses of RO4929097 of 80mg (cohort 1) or recommended Phase II dose (cohort 2) on a 3 days on 4 days off schedule. Anticipated time on study treatment is until disease progression or unacceptable toxicity. Target sample size is <50.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >/= 18 years of age
* stage IIIB/IV recurrent or refractory non-small cell lung cancer
* at most 2 lines of prior therapy in the metastatic setting (first line: platinum containing regimen and bevacizumab; second line: EGFR-targeted therapy)
* ECOG performance status 0-2
* adequate liver, renal and bone marrow function

Exclusion Criteria:

* prior chemotherapy or radiotherapy </= 4 weeks before first dose of study drug
* history of other malignancy within the past 2 years, except for basal cell skin carcinoma or in situ cervical carcinoma
* history of CNS metastases or leptomeningeal metastases, except for clinically stable disease
* serious cardiovascular illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2010-01; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Tumour blood flow and tumour metabolic response rate | PET and CT assessments on day 4 (cycle 1) and day 16 (cycles 1 and 2)

SECONDARY OUTCOMES:
Pharmacokinetic profile and pharmacodynamic parameters (e.g. changes in circulating endothelial and hematopoietic precursors) | pharmacokinetics: cycle 1 on days 1, 2, 4, 10, 11, 16; cycle 2 on days 1, 2, 16\npharmacodynamics: cycle 1 on days 1, 2, 4, 11, 16; cycle 2 on days 1, 16
Tumour response according to RECIST criteria | assessments once every 2nd cycle on day 16
Safety and tolerability: AEs, laboratory parameters | throughout study, laboratory assessments on days 1, 8 and 15 of each cycle

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Amsterdam, Netherlands